CLINICAL TRIAL: NCT01104259
Title: Phase I Study of ABT-888 in Combination With Cisplatin and Vinorelbine for Patients With Advanced Triple Negative Breast Cancer and/or BRCA-Mutation Associated Breast Cancer
Brief Title: Veliparib, Cisplatin, and Vinorelbine Ditartrate in Treating Patients With Recurrent and/or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7161; NCI-2010-00356 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH); 7161 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium)
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Estrogen Receptor-negative Breast Cancer; HER2-negative Breast Cancer; Hereditary Breast/Ovarian Cancer - BRCA1; Hereditary Breast/Ovarian Cancer - BRCA2; Male Breast Cancer; Progesterone Receptor-negative Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer; Triple-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — veliparib; Cisplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (veliparib with cisplatin and vinorelbine tartrate) (Experimental): Patients receive veliparib PO BID on days 1-14 (days 0-13 of course 1 only). Patients also receive cisplatin IV over 1 hour on day 1 and vinorelbine ditartrate IV over 10-20 minutes on days 1 and 8. Treatment repeats every 21 days for 6-10 courses in the absence of disease progression or unacceptable toxicity. Treatment with veliparib alone may continue in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: veliparib; Drug: cisplatin; Drug: vinorelbine tartrate; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: veliparib — Given PO
  Other Names: ABT-888
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: vinorelbine tartrate — Given IV
  Other Names: Eunades; navelbine ditartrate; NVB; VNB
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of veliparib when given together with cisplatin and vinorelbine ditartrate in treating patients with breast cancer that has returned or spread to other parts of the body. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin and vinorelbine ditartrate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving veliparib together with combination chemotherapy may be a better treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of ABT-888 (veliparib) when administered daily for 14 days out of a 21 day cycle in combination with cisplatin and vinorelbine (vinorelbine ditartrate) in subjects with metastatic triple negative breast cancer (TNBC) and breast cancer (BRCA) mutation associated breast cancer.

SECONDARY OBJECTIVES:

I. Assess the pharmacokinetic profile of ABT-888 when combined with cisplatin and vinorelbine and the safety/tolerability profile of the combination.

II. Evaluate the level of poly ADP ribose polymerase (PARP) inhibition at each dose level to determine whether maximal PARP inhibition is achieved.

III. Identify the subgroup of triple negative breast cancer patients who will potentially derive the most benefits from PARP inhibition combined with platinum-based chemotherapy.

OUTLINE: This is a dose-escalation study of veliparib.

Patients receive veliparib orally (PO) twice daily (BID) on days 1-14 (days 0-13 of course 1 only). Patients also receive cisplatin intravenously (IV) over 1 hour on day 1 and vinorelbine ditartrate IV over 10-20 minutes on days 1 and 8. Treatment repeats every 21 days for 6-10 courses in the absence of disease progression or unacceptable toxicity. Treatment with veliparib alone may continue in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent and/or metastatic breast cancer
* Subjects must meet at least one of the following two criteria:

  * Histologically confirmed primary or metastatic site that is estrogen receptor (ER)-negative (less than 10%), progesterone receptor (PR)-negative (less than 10%), and human epidermal growth factor receptor (HER)2 non-over expressing by immunohistochemistry (IHC) (0, 1) or non-amplified by fluorescence in situ hybridization (FISH)
  * Confirmed BRCA1 or BRCA2 mutation associated breast cancer
* Subjects must have measurable disease, defined as at least one lesion that can be measured in at least one dimension with a minimum size of: longest diameter >= 10 mm (computed tomography [CT] scan slice thickness no greater than 5 mm); 10 mm caliper measurement by clinical exam; to be considered pathologically enlarged and measurable, a lymph node must be >= 15 mm in short axis when assessed by CT scan
* Subjects may have had any number of prior chemotherapy, endocrine therapy, immunologic, or biologic regimens for metastatic breast cancer
* Performance status >= 60% on the Karnofsky scale (Eastern Cooperative Oncology Group [ECOG] =< 2)
* Absolute neutrophil count (ANC) >= 1,500/mm^3 (1.5 x 10^9/L)
* Platelets >= 100,000/mm^3 (100 x 10^9/L)
* Hemoglobin >= 9.0 g/dL
* Serum creatinine =< 1.5 x upper normal limit of institution's normal range OR creatinine clearance >= 50 mL/min/1.73 m^2 for subjects with creatinine levels above institutional normal
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 2.5 x the upper normal limit of institution's normal range; for subjects with liver metastases, AST and/or ALT < 5 x the upper normal limit of institution's normal range
* Bilirubin =< 1.5 x the upper normal limit of institution's normal range; subjects with Gilbert's syndrome may have a bilirubin > 1.5 x the upper normal limit of institution's normal range
* Partial thromboplastin time (PTT) must be =< 1.5 x the upper normal limit of institution's normal range and international normalized ratio (INR) < 1.5; subjects on anticoagulant (such as Coumadin) will have PTT and INR as determined by the investigator
* Women of childbearing potential must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and for 90 days following completion of therapy; women of childbearing potential must have a negative serum pregnancy test within 21 days prior to initiation of treatment and/or be confirmed as having postmenopausal status; criteria for determining menopause include any of the following: prior bilateral oophorectomy; age >= 60 years; age < 60 years and amenorrheic for at least 12 months in the absence of chemotherapy, endocrine therapy, or ovarian suppression and follicle-stimulating hormone (FSH) and estradiol in the postmenopausal range;

  * Total abstinence from sexual intercourse (minimum one complete menstrual cycle)
  * Vasectomized partner of female subjects
  * Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration
  * Double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream)
  * Intra-uterine device (IUD)
* Male subjects (including those who are vasectomized) whose partners are pregnant or might be pregnant must agree to use condoms for the duration of the study and for 90 days following completion of therapy
* Radiation therapy of a non-target lesion must have been completed at least 2 weeks prior to the enrollment date
* Subjects with known brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 14 days of stable neurologic function prior to the first dose of study drug
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subject has received any anti-cancer therapy including chemotherapy, immunotherapy, biologic or any investigational therapy within either 28 days or 5 half-lives of a targeted therapy (whichever is shorter), prior to study drug administration; subjects receiving hormone therapy, bisphosphonates, denosumab or luteinizing-hormone-releasing hormone (LHRH)-agonists are eligible; subjects who have not recovered to within one grade level (not to exceed grade 2) of their baseline following a significant adverse event or toxicity attributed to prior anti-cancer treatment are excluded
* Subjects with a known hypersensitivity to platinum compounds or vinorelbine
* Subjects with baseline peripheral neuropathy that exceeds grade 1
* Clinically significant and uncontrolled major medical condition(s) including but not limited to:

  * Active uncontrolled infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris or cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements
  * Any medical condition, which in the opinion of the study investigator, places the subject at an unacceptably high risk for toxicities
  * Subjects with significant fluid retention, including ascites or pleural effusion, may be allowed at the discretion of the principal investigator
* Subject is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
MTD of veliparib, defined as the highest dose tested in which fewer than 33% of patients experienced dose-limiting toxicity attributable to the study regimen, when at least 6 patients were treated at that dose and were evaluable for toxicity | Day 21

SECONDARY OUTCOMES:
Toxicity profile, defined by the incidence of toxicity, as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days post-treatment
Pharmacokinetic (PK) parameters of veliparib in plasma and urine samples | Baseline and day 1 of courses 1 and 4
  The PK parameters determined will be: AUC0-t (the area under the concentration-time curve over a dosing interval), Cmax (maximal concentration), Tmax (time to maximal concentration), Vd (volume of distribution), CL/F (oral clearance for veliparib), CL (clearance for cisplatin), and t1/2 (elimination half-life). To improve understanding of systemic bioavailability, the amount of veliparib excreted in the urine for each collection interval will be calculated by the product of urinary drug concentration and urine volume.
Pharmacokinetic (PK) parameters of cisplatin in plasma samples | Baseline and day 1 of courses 1 and 4
  The PK parameters determined will be: AUC0-t, Cmax, Tmax, Vd, CL/F, CL, and t1/2 .
Pharmacodynamic parameters of PARP inhibition | Baseline and day 1 of courses 1 and 4
  Assessed by measuring changes in PAR levels in peripheral blood mononuclear cells and in tumor tissue (if available).

OTHER OUTCOMES:
Progression-free survival | The number of days from the date the subject started study drug to the date the subject experiences an event of disease progression, or to the date of death if disease progression is not reached, assessed up to 30 days
  Estimated using Kaplan-Meier methodology and 95% confidence interval.
Time to disease progression | The number of days from the date the subject started study drug to the date of the subject's disease progression, assessed up to 30 days
  Estimated using Kaplan-Meier methodology and 95% confidence interval.
Proportion of patients achieving a complete response (CR) or partial response (PR) (objective response rate) | Up to 30 days
  Assessed by Response Evaluation Criteria in Solid Tumors version 1.1 and estimated with 95% confidence interval.
Duration of overall response | The number of days from the day the criteria are met for CR or PR (whichever is recorded first) to the date that progressive disease is objectively documented, assessed up to 30 days
  Estimated using Kaplan-Meier Methodology.
ECOG performance status | Up to 30 days
  Descriptive statistics will be summarized for each assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Specht, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States